CLINICAL TRIAL: NCT06078592
Title: Comparison of Efficacy and Ocular Surface Disease Assessment Between BRIDIN- PLUS® Eye Drops and COMBIGAN® Eye Drops in Glaucoma or Ocular Hypertensive Patients
Brief Title: Comparison of Efficacy and Ocular Surface Assessment Between BRIDIN-plus and Combigan in Glaucoma or Ocular Hypertensive
Acronym: BCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHA University (Other)
Collaborators: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BCT
Record Dates: First submitted 2023-07-19; First posted 2023-10-12 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Glaucoma; Ocular Hypertensive
MeSH Terms: conditions — Glaucoma | interventions — Brimonidine Tartrate; Timolol; Preservatives, Pharmaceutical

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRIDIN-plus Eye drops (Experimental): One drop in the eyes, twice a day, approximately 12 hours apart.
  Interventions: Drug: BRIDIN-plus Eye drops
- Combigan Eye drops (Active Comparator): One drop in the eyes, twice a day, approximately 12 hours apart.
  Interventions: Drug: Combigan Eye drops

INTERVENTIONS:
Drug: BRIDIN-plus Eye drops — BRIDIN-plus Eye drops
  Other Names: Brimonidine tartrate 2.0mg, Timolol maleate 6.8mg(without preservative)
  Arms: BRIDIN-plus Eye drops
Drug: Combigan Eye drops — Combigan Eye drops
  Other Names: Brimonidine tartrate 2.0mg, Timolol maleate 6.8mg(with preservative)
  Arms: Combigan Eye drops

SUMMARY:
Comparison of Efficacy and Ocular Surface Disease Assessment between BRIDIN-plus Eye drops and Combigan Eye drops in Glaucoma or Ocular Hypertensive Patients : Phase 4, Parallel Group Design, Investigator-blind, Active-control, Randomized, Multi-center Trial

DETAILED DESCRIPTION:
The purpose of this clinical trial is to prove lower negative effects on ocular surface disease and higher patient compliance of a single-use formula BRIDIN-PLUS® eye drops group, comparing to a multi-use formula COMBIGAN® eye drops after 12 weeks of administration to glaucoma or ocular hypertensive patients.

ELIGIBILITY:
Inclusion Criteria

1. Male or female adults who are 19 years or older with a diagnosis of glaucoma or intraocular hypertension
2. A person who has completed an appropriate washout period if glaucoma treatment medication has been used
3. Intraocular pressure measured by Goldman applanation tonometer at visit 2 is 15mmHg or above and less than 40mmHg
4. A person who has signed the written consent form by himself/herself or by a legal representative

Exclusion Criteria:

1. A patient with primary close angle glaucoma, congenital glaucoma, secondary glaucoma caused by steroids
2. Best corrected visual acuity of both eyes measured by Snellen acuity charts is 20/80 (decimal 0.25) or less
3. A patient with progressive intraocular inflammation
4. Central corneal thickness is less than 470um or greater than 591ums
5. A patient who has had lacrimal punctual occlusion done within the last 3 monthds or who has eye surgery plan during the clinical study
6. Pregnant or lactating women
7. Other cases if investigators judge the patient is difficult to participate the clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Corneal staining test | 12 weeks after administration
  Corneal staining score is evaluated according to the oxford grading system after blue fluorescein staining under a slit lamp biomicroscope of cobalt blue light source using a yellow filter. Corneal surface is divided into 3 areas and evaluated from grade 0 indicating that there is no staining to grade 5 indicating denser staining due to severe corneal defect. (The score ranges from 0 to 5, with higher scores indicate worse symtoms.)
Conjunctival staining test | 12 weeks after administration
  Conjunctival staining score is evaluated after blue fluorescein staining under a slit lamp biomicroscope, by NEI(The National Eye Institute) scale. Conjunctival surface is divided into 6 areas and evaluated from grade 0 indicating that there is no staining to grade 3 indicating denser staining due to severe conjunctival defect.
Ocular surface disease index (OSDI) | 12 weeks after administration
  Ocular surface disease index include 12 items comprising of assessment of vision related functioning (5 items), ocular symptoms(4 items) and environmental factors that may cause symptoms (3 items). Each item is 5-point Likert scale in which a higher score indicates more severe symptoms.
  A total score is classified as normal (0-12), mild (13-22), moderate (23-32) and severe (33 or more) and it is evaluated based on grades and score changes
Questionnaire (Evaluation of Satisfaction with Medication, Ocular tolerance) | 12 weeks after administration
  treatment administration satisfaction and ocular tolerance are evaluated through questionnaires. Treatment administration satisfaction questionnaire includes the convenience of use and storage of investigational products and ocular tolerance evaluation questionnaire includes symptom severity(0~3) and symptom duration(briefly, persistent) for 8 symptoms of stinging/burning, sticky eyes, itching, blurred vision, foreign-body sensation, dryness, photophobia, pain. Medication compliance is evaluated with MGL-MAQ-Korean version.

SECONDARY OUTCOMES:
Corneal staining test | 4 weeks after administration
  Corneal staining score is evaluated according to the oxford grading system after blue fluorescein staining under a slit lamp biomicroscope of cobalt blue light source using a yellow filter. Corneal surface is divided into 3 areas and evaluated from grade 0 indicating that there is no staining to grade 5 indicating denser staining due to severe corneal defect. (The score ranges from 0 to 5, with higher scores indicate worse symtoms.)
Conjunctival staining test | 4 weeks after administration
  Conjunctival staining score is evaluated after blue fluorescein staining under a slit lamp biomicroscope, by NEI(The National Eye Institute) scale. Conjunctival surface is divided into 6 areas and evaluated from grade 0 indicating that there is no staining to grade 3 indicating denser staining due to severe conjunctival defect.
Ocular surface disease index (OSDI) | 4 weeks after administration
  Ocular surface disease index include 12 items comprising of assessment of vision related functioning (5 items), ocular symptoms(4 items) and environmental factors that may cause symptoms (3 items). Each item is 5-point Likert scale in which a higher score indicates more severe symptoms.
  A total score is classified as normal (0-12), mild (13-22), moderate (23-32) and severe (33 or more) and it is evaluated based on grades and score changes
IOP(Intraocular pressure) | 4, 12 weeks after administration
  The same tonometer (Goldman applanation tonometer) should be used. In the case of bilateral glaucoma, intraocular pressure of the right eye is first measured and a higher one is used. If intraocular pressures of both eyes are the same, intraocular pressures of the right eye is used. In unilateral glaucoma, intraocular pressures of an eye with glaucoma is used.
Tear break up time (TBUT) | 4, 12 weeks after administration
  Corneal staining score is evaluated after blue fluorescein staining on a 6-point scale according to oxford grading system under a slit lamp biomicroscope with a yellow filter offering cobalt blue light. After blue fluorescein staining, a participant is asked to blink their eyes. Then, time from the last blinking to the point when black spots, lines or loss of fluorescein are observed is measured in seconds under a slit lamp biomicroscope with a yellow filter offering cobalt blue light. The mean value of three repeated measurement results are used
Hyperemia score | 4, 12 weeks after administration
  Prior to fluorescein staining, hyperemia evaluation is done to the bulbar conjunctiva and the limbus, the border between cornea and conjunctiva using Efron Grading Scales. grade 0: normal; grade 1: trace; grade 2: mild; grade 3: moderate; grade 4: severe (The scales from grade 0 to 4, with higer scales indicate greater severity of symptoms.)

CONTACTS AND LOCATIONS:
Overall Officials: Seungsoo Rho, MD, PhD, Principal Investigator — CHA Bundang Medical Center
Locations (1):
- Seungsoo Rho, Seoul, Seongnam, Bundang-gu, South Korea